CLINICAL TRIAL: NCT03722264
Title: An Evaluation of Protective Effects of OpalSeal™ Against Early Dental Decay in Orthodontic Patients. A Pilot Study
Brief Title: An Evaluation of Protective Effects of OpalSeal™ Against Early Dental Decay in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: HM20011025
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Results first posted 2020-02-25 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Cavities of Teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Participants have at least two teeth planned for extraction on either side of the mouth. The study will use a split-mouth design with random assignments for intervention (OpalSeal) on one tooth.
Who Masked: Participant, Outcomes Assessor
Masking Description: Opalseal and TransbondXT are identical in color, consistency and application allowing random assignments as well as patient blinding.
  The outcomes assessor will also be blinded to the groups assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- OpalSeal (Experimental): OpalSeal will be applied
  1. to the buccal surfaces of to-be-extracted teeth on one side of the mouth which will be determined randomly for each participant during bonding of orthodontic brackets, or
  2. to the proximal surfaces following IPR in accordance to manufacturer instructions. Since OpalSeal has fluoride releasing capability, this would be experimental arm
  Interventions: Device: OpalSeal
- Transbond XT (Placebo Comparator): TransbondXT will be applied
  1. to the buccal surfaces of to-be-extracted teeth on the other side of the mouth which will be determined based on which side received OpalSeal for each participant during bonding of orthodontic brackets, or
  2. to the proximal surfaces following IPR in accordance to manufacturer instructions. Transbond XT does not have fluoride and hence would be considered as a placebo.
  Interventions: Device: TransbondXT

INTERVENTIONS:
Device: OpalSeal — OpalSeal is a fluoride releasing orthodontic primer that is FDA approved for use during bonding of orthodontic brackets
  Arms: OpalSeal
Device: TransbondXT — Transbond is a primer used to bond orthodontic brackets that does not contain fluoride
  Arms: Transbond XT

SUMMARY:
Fluoride is very effective in preventing dental decay (cavities) when applied in the form of a varnish on tooth surfaces. The purpose of this study is to verify if fluoride-releasing primer (OpalSeal) offers more protection against early dental decay (cavity) compared to conventional primer (Transbond XT) during treatment with braces.

DETAILED DESCRIPTION:
Primers are a type of 'glue' routinely used in orthodontics to attach brackets (metallic components) to the teeth. OpalSeal is a fluoride-releasing primer that has the potential to reduce cavities in patients receiving braces.

Orthodontic patients are at particular risk of developing two types of early carious lesions (decay):

1. Around the brackets called White Spot Lesions and
2. Along the sides of the teeth after slenderization procedure called inter-proximal reduction (IPR).

Our research questions are:

1. Can OpalSeal offer protection against white spot lesions (WSL) around the brackets?
2. Can OpalSeal offer protection against decay on the sides of teeth following IPR?

ELIGIBILITY:
Inclusion Criteria:

* Patients age 10 and older seeking treatment at the VCU Orthodontics Clinic who require extraction of at least 2 teeth for orthodontic purposes
* Such teeth should be free of any developmental defects

Exclusion Criteria:

* Patients under 10 years of age
* Patients with defective teeth
* Those who cannot provide consent/assent OR not able to follow research protocols
* Protected population (prisoners)

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parthasarathy Madurantakam, DDS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- School of Dentistry, Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 participants were enrolled with all participants receiving each treatment
Groups:
- Bilateral Treatment With OpalSeal and Transbond XT: Experimental: OpalSeal OpalSeal will be applied
  to the buccal surfaces of to-be-extracted teeth on one side of the mouth which will be determined randomly for each participant during bonding of orthodontic brackets, or to the proximal surfaces following IPR in accordance to manufacturer instructions. Since OpalSeal has fluoride releasing capability, this would be experimental arm.
  Placebo Comparator: Transbond XT TransbondXT will be applied
  to the buccal surfaces of to-be-extracted teeth on the other side of the mouth which will be determined based on which side received OpalSeal for each participant during bonding of orthodontic brackets, or to the proximal surfaces following IPR in accordance to manufacturer instructions. Transbond XT does not have fluoride and hence would be considered as a placebo.
Period: Overall Study
Arm/Group | Bilateral Treatment With OpalSeal and Transbond XT
Started | 12
Completed | 9
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: Although age was used to determine inclusion/exclusion into the study, data on age was not stored after enrollment.
  Gender, and race/ethnicity data was not collected as they are not relevant variables for the outcomes studied
Arm/Group | Bilateral Treatment With OpalSeal and Transbond XT
Number analyzed (Participants) | 9
Age, Customized [Count of Participants; unit: Participants] | NA — Data not stored after enrollment
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex not measured | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Loss of Mineral Density in the Enamel
Description: Teeth will be subjected to microCT to assess the extent of demineralization. Loss of mineral density will be measured as depth of lesions
Time Frame: Time from initial bonding to extraction (max 90 days)
Population: 9 teeth in each group were available for analysis
Measure: Mean (Full Range); unit: microns
Units Other Than Participants: teeth
Groups:
- OpalSeal: OpalSeal will be applied
  1. to the buccal surfaces of to-be-extracted teeth during bonding of orthodontic brackets, or
  2. to the proximal surfaces following IPR in accordance to manufacturer instructions. Since OpalSeal has fluoride releasing capability, this would be experimental arm,
  OpalSeal: OpalSeal is a fluoride releasing orthodontic primer that is FDA approved for use during bonding of orthodontic brackets
- Transbond XT: TransbondXT will be applied
  1. to the buccal surfaces of to-be-extracted teeth during bonding of orthodontic brackets, or
  2. to the proximal surfaces following IPR in accordance to manufacturer instructions. Transbond XT does not have fluoride and hence would be considered as a placebo.
  TransbondXT: Transbond is a primer used to bond orthodontic brackets that does not contain fluoride
Arm/Group | OpalSeal | Transbond XT
Number analyzed (Participants) | 9 | 9
Number analyzed (teeth) | 9 | 9
microns | 70.8 [0 to 130.5] | 77.4 [0 to 245.3]

2. Secondary Outcome: Surface Topography and Hardness
Description: Scanning electron microscopy and atomic force microscopy will be used to evaluate the protective effect of OpalSeal
Time Frame: Time from initial bonding to extraction (max 90 days)
Population: Data could not be collected for this variable.
Arm/Group | OpalSeal | Transbond XT
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Retention of OpalSeal
Description: The protective effects of OpalSeal is subject to its retention at the site of application. Since OpalSeal fluoresces under black light, its retention will be evaluated
Time Frame: Time from initial bonding to extraction (max 90 days)
Population: TransbondXT retention cannot be assessed so no control teeth were analyzed. Only 5 teeth on which OpalSeal was applied were analyzed
Measure: Median (Full Range); unit: percent coverage
Arm/Group | OpalSeal | Transbond XT
Number analyzed (Participants) | 5 | 0
percent coverage | 28.1 [0 to 37.5] |

ADVERSE EVENTS:
Time Frame: The study looked at participant teeth in an orthodontic setting. No medical data, including untoward or unfavorable medical occurrences, about the participants was available or collected for the study.
Description: The study looked at participant teeth in an orthodontic setting. No medical data, including untoward or unfavorable medical occurrences, about the participants was available or collected for the study.
Arm/Group | OpalSeal | Transbond XT
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT03722264/Prot_001.pdf